CLINICAL TRIAL: NCT03173248
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of AG-120 in Combination With Azacitidine in Subjects ≥ 18 Years of Age With Previously Untreated Acute Myeloid Leukemia With an IDH1 Mutation
Brief Title: Study of AG-120 (Ivosidenib) vs. Placebo in Combination With Azacitidine in Participants With Previously Untreated Acute Myeloid Leukemia With an IDH1 Mutation
Acronym: AGILE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG120-C-009
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Newly Diagnosed Acute Myeloid Leukemia (AML); Untreated AML; AML Arising From Myelodysplastic Syndrome (MDS); Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Leukemia; Azacitidine; AG-120; ivosidenib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — ivosidenib; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG-120 + Azacitidine (Experimental): Participants received AG-120 500 mg orally, once daily (QD) in combination with azacitidine 75 milligrams per square meter per day (mg/m^2/day) subcutaneously (SC) or intravenously (IV), on Days 1-7, or on Days 1-5 and 8-9, of each 28-day cycle for a minimum of 6 cycles until death, disease relapse, disease progression, development of unacceptable toxicity (adverse event), confirmed pregnancy, withdrawal by participant or protocol violation.
  Interventions: Drug: AG-120; Drug: Azacitidine
- Placebo + Azacitidine (Placebo Comparator): Participants received AG-120 matching placebo orally, QD in combination with azacitidine 75 mg/m^2/day SC or IV, on Days 1-7, or on Days 1-5 and 8-9, of each 28-day cycle for a minimum of 6 cycles until death, disease relapse, disease progression, development of unacceptable toxicity (adverse event), confirmed pregnancy, withdrawal by participant or protocol violation .
  Interventions: Drug: Placebo; Drug: Azacitidine

INTERVENTIONS:
Drug: AG-120 — Tablets administered orally
  Other Names: Ivosidenib
  Arms: AG-120 + Azacitidine
Drug: Placebo — Tablets administered orally
  Arms: Placebo + Azacitidine
Drug: Azacitidine — Administered SC or IV
  Other Names: Vidaza®

SUMMARY:
Study AG120-C-009 is a global, Phase 3, multicenter, double-blind, randomized, placebo-controlled clinical trial to evaluate the efficacy and safety of AG-120 (ivosidenib) + azacitidine vs placebo + azacitidine in adult participants with previously untreated IDH1m AML who are considered appropriate candidates for non-intensive therapy. The primary endpoint is event-free survival (EFS). The key secondary efficacy endpoints are overall survival (OS), rate of complete remission (CR), rate of CR and complete remission with partial hematologic recovery (CRh), and overall response rate (ORR). Participants eligible for study treatment based on Screening assessments will be randomized 1:1 to receive oral AG-120 or matched placebo, both administered in combination with subcutaneous (SC) or intravenous (IV) azacitidine. An estimated 200 participants will take part in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age and meet at least 1 of the following criteria defining ineligibility for intensive induction chemotherapy (IC): ≥ 75 years old, Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 2, severe cardiac disorder (e.g., congestive heart failure requiring treatment, left ventricular ejection fraction (LVEF), ≤50%, or chronic stable angina), severe pulmonary disorder (e.g., diffusing capacity of the lungs for carbon monoxide ≤65% or forced expiratory volume in 1 second ≤65%), creatinine clearance <45 mL/minute, bilirubin >1.5 times the upper limit of normal (ULN) and/or have any other comorbidity that the Investigator judges to be incompatible with intensive IC and must be reviewed and approved by the Medical Monitor before study enrollment.
2. Have previously untreated AML, defined according to World Health Organization (WHO) criteria, with ≥ 20% leukemic blasts in the bone marrow. Participants with extramedullary disease alone (i.e., no detectable bone marrow and no detectable peripheral blood AML) are not eligible for the study.
3. Have an isocitrate dehydrogenase 1 (IDH1) mutation.
4. Have an ECOG PS score of 0 to 2.
5. Have adequate hepatic function.
6. Have adequate renal function.
7. Have agreed to undergo serial blood and bone marrow sampling.
8. Be able to understand and willing to sign an informed consent form (ICF).
9. Be willing to complete Quality of Life assessments during the study
10. If female with reproductive potential, must have a negative serum pregnancy test prior to the start of study therapy. Females of reproductive potential, as well as fertile men and their female partners of reproductive potential, must agree to use 2 effective forms of contraception.

Exclusion Criteria:

1. Are candidates for and willing to receive intensive induction chemotherapy (IC) for their AML.
2. Have received any prior treatment for AML with the exception of hydroxyurea.
3. Have received a hypomethylating agent for myelodysplastic syndrome (MDS).
4. Participants who had previously received an experimental agent for MDS may not be randomized until a washout period has elapsed since the last dose of that agent.
5. Have received prior treatment with an IDH1 inhibitor.
6. Have a known hypersensitivity to any of the components of AG-120, matched placebo, or azacitidine.
7. Are female and pregnant or breastfeeding.
8. Have an active, uncontrolled, systemic fungal, bacterial, or viral infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
9. Have a prior history of cancer other than MDS or myeloproliferative disorder, unless the participant has been free of the disease for ≥ 1 year prior to the start of study treatment.
10. Have had significant active cardiac disease within 6 months prior to the start of the study treatment.
11. Have any condition that increases the risk of abnormal ECG or cardiac arrhythmia.
12. Have a condition that limits the ingestion or absorption of drugs administered by mouth.
13. Have uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg).
14. Have clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia.
15. Have immediate, life-threatening, severe complications of leukemia, such as uncontrolled bleeding, pneumonia with hypoxia or sepsis, and/or disseminated intravascular coagulation.
16. Have any other medical or psychological condition deemed by the Investigator to be likely to interfere with the participant's ability to give informed consent or participate in the study.
17. Are taking medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥5 half-lives prior to dosing, or unless the medications can be properly monitored during the study. (If equivalent medication is not available, heart rate corrected QT interval [QTc] will be closely monitored.)
18. Have a known medical history of progressive multifocal leukoencephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (2):
  - Norton Cancer Institute - Suburban, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
- Austria (2):
  - Salzburger Landeskliniken, Salzburg
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhugel, Vienna
- Brazil (6):
  - Unicamp Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
  - Hospital Sao Jose, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Canada (2):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - University Health Network, Toronto, Ontario
- China (6):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
- Fakultni nemocnice Ostrava, Ostrava, Czechia
- France (14):
  - Hopital Haut Leveque, Pessac, Gironde
  - Hopital Bretonneau, Tours, Indre-et-Loire
  - Hotel Dieu - Nantes, Nantes, Loire-Atlantique
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - CHRU de Brest - Hopital Morvan, Brest
  - Institut dHematologie de Basse Normandie, Caen
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier de Versailles CHV Hopital Andre Mignot, Le Chesnay
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - CHRU de Poitiers La Miletrie, Poitiers
  - Hopital de Hautepierre, Strasbourg
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Charite - Universitatsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - LMU Klinikum der Universitat Munchen, München
  - Universitatsklinikum Ulm, Ulm
- Israel (3):
  - Rabin Medical Center - PPDS, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Shamir Medical Center Assaf Harofeh, Tzrifin
- Italy (7):
  - ASST dei Sette Laghi - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Ospedale Infermi di Rimini, Rimini
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (4):
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - University of Fukui Hospital, Fukui
  - Japanese Red Cross Society Himeji Hospital, Himeji
  - Kobe City Medical Center General Hospital, Kobe
- Mexico (2):
  - SINACOR, Culiacán
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen, Nijmegen
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
- Russia (2):
  - Kaluga Regional Clinical Hospital, Kaluga
  - City Clinical Hospital # 40, Moscow
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Pusan National University Hospital, Busan
  - Severance Hospital Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
- Spain (13):
  - CHUS H. Clinico U. de Santiago, Santiago de Compostela, A Coruna
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (5):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
- Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Montesinos P, Recher C, Vives S, Zarzycka E, Wang J, Bertani G, Heuser M, Calado RT, Schuh AC, Yeh SP, Daigle SR, Hui J, Pandya SS, Gianolio DA, de Botton S, Dohner H. Ivosidenib and Azacitidine in IDH1-Mutated Acute Myeloid Leukemia. N Engl J Med. 2022 Apr 21;386(16):1519-1531. doi: 10.1056/NEJMoa2117344. PMID 35443108
- [Derived] Montesinos P, Marchione DM, Recher C, Heuser M, Vives S, Zarzycka E, Wang J, Riva M, Calado RT, Schuh AC, Yeh SP, Tron AE, Hui J, Gianolio DA, Choe S, Patel P, De Botton S, DiNardo CD, Dohner H. Long-term results from the AGILE study of azacitidine plus ivosidenib vs placebo in newly diagnosed IDH1-mutated AML. Blood Adv. 2025 Oct 28;9(20):5177-5189. doi: 10.1182/bloodadvances.2025016399. PMID 40706052
- [Derived] Woods A, Norsworthy KJ, Wang X, Vallejo J, Chiu Yuen Chow E, Li RJ, Sun J, Charlab R, Jiang X, Pazdur R, Theoret MR, de Claro RA. FDA Approval Summary: Ivosidenib in Combination with Azacitidine for Treatment of Patients with Newly Diagnosed Acute Myeloid Leukemia with an IDH1 Mutation. Clin Cancer Res. 2024 Apr 1;30(7):1226-1231. doi: 10.1158/1078-0432.CCR-23-2234. PMID 38010220
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 199 investigational sites from 19 March 2018 to 18 March 2021 (data cut off date). This study is ongoing. Results collected through data cut off date, 18 March 2021 are being reported.
Pre-assignment Details: A total of 146 participants with previously untreated isocitrate dehydrogenase 1 mutation-positive (IDH1m) acute myeloid leukemia (AML) were randomized into a 1:1 ratio to receive ivosidenib (AG-120) or AG-120 matched placebo in combination with azacitidine.
Groups:
- Placebo + Azacitidine: Participants received AG-120 matching placebo orally, QD in combination with azacitidine 75 mg/m^2/day SC or IV, on Days 1-7, or on Days 1-5 and 8-9, of each 28-day cycle for a minimum of 6 cycles until death, disease relapse, disease progression, development of unacceptable toxicity (adverse event), confirmed pregnancy, withdrawal by participant or protocol violation.
Period: Overall Study
Arm/Group | AG-120 + Azacitidine | Placebo + Azacitidine
Started | 72 | 74
Safety Analysis Set (Safety Analysis Set (SAS) included all participants who received at least 1 dose of the study treatment.) | 71 | 73
Completed | 0 | 0
Not Completed | 72 | 74
Not completed — Death | 28 | 46
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Ongoing at Data Cut-off Date: 18 March 2021 | 38 | 23

BASELINE CHARACTERISTICS:
Population: FAS included all participants who were randomized.
Groups:
- AG-120 + Azacitidine: Participants received AG-120 500 mg orally, QD in combination with azacitidine 75 mg/m^2/day SC or IV, on Days 1-7, or on Days 1-5 and 8-9, of each 28-day cycle for a minimum of 6 cycles until death, disease relapse, disease progression, development of unacceptable toxicity (adverse event), confirmed pregnancy, withdrawal by participant or protocol violation.
- Total: Total of all reporting groups
Arm/Group | AG-120 + Azacitidine | Placebo + Azacitidine | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (6.18) | 75.2 (7.39) | 74.8 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 42 | 38 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 21 | 32 | 53
  Unknown or Not Reported | 45 | 41 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 15 | 19 | 34
  Race: White | 12 | 12 | 24
  Race: Black or African American | 0 | 2 | 2
  Race: Other | 1 | 1 | 2
  Race: Not Reported | 44 | 40 | 84

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from randomization until treatment failure, relapse from remission, or death from any cause, whichever occurs first. Treatment failure was defined as failure to achieve complete remission (CR) by Week 24. CR: Bone marrow blasts <5% and no Auer rods; absence of extramedullary disease; Absolute neutrophil count (ANC) ≥1.0 × 10^9 per litre (10^9/L) (1000 per microlitre [1000/μL]); platelet count ≥100 × 10^9/L (100,000/μL); independence of red blood cell transfusions. Participants who had an EFS event (relapse or death) after, 2 or more missing disease assessments were censored at the last adequate disease assessment documenting no relapse before the missing assessments. The reported data represents the Kaplan-Meier median value.
Time Frame: Up to Week 24
Population: FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 72 | 74
months | 0.03 [0.03 to 11.01] | 0.03 [NA to NA] — The upper and lower limit of 95% confidence interval (CI) were not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: AG-120 + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.0011, Log Rank — P-value is calculated from the one-sided log-rank test stratified by the randomization stratification factors (AML status and geographic region); Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.16 to 0.69] — Hazard ratio is estimated using a Cox's proportional hazards model stratified by the randomization stratification factors (AML status and geographic region) with placebo + azacitidine as the denominator

2. Secondary Outcome: Complete Remission Rate (CR Rate)
Description: CR rate is defined as the proportion of participants who achieve a CR. A Cochran-Mantel-Haenszel (CMH) test will be used to compare CR rate between the 2 treatment arms.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to the date of death due to any cause. Kaplan-Meier (KM) curves and KM estimates of OS will be presented for each treatment arm.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

4. Secondary Outcome: CR + Complete Remission With Partial Hematologic (CRh) Rate
Description: CR + CRh rate is defined as the proportion of participants who achieve a CR or CRh. CRh is defined as a CR with partial recovery of peripheral blood counts (less than 5% bone marrow blasts, absolute neutrophil count (ANC) greater than 0.5 × 10^9/liter (L) 500/microliter (μL)], and platelets greater than 50 × 10^9/L [50,000/μL]). A CMH test will be used to compare the CR + CRh rate between the 2 treatment arms.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the rate of CR, CR with incomplete hematologic recovery (CRi) (including CR with incomplete platelet recovery [CRp]), partial remission (PR), and morphologic leukemia-free state (MLFS). The best response is calculated using the following hierarchy: CR, followed by CRi (including CRp), followed by PR and MLFS. A summary of best response by treatment arm will be produced. A CMH test will be used to compare ORR between the 2 treatment arms.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

6. Secondary Outcome: CR + CRi (Including CRp) Rate
Description: The CR + CRi (including CRp) rate is defined as the proportion of participants who achieve a CR or CRi (including CRp). A CMH test will be used to compare the CR + CRi (including CRp) rate between the 2 treatment arms.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

7. Secondary Outcome: Duration of CR (DOCR)
Description: DOCR will be calculated as the date of the first occurrence of CR to the date of first documented disease relapse, or death. DOCR is only defined for participants who achieve a CR.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Duration of CRh (DOCRh)
Description: DOCRh will be calculated as the date of the first occurrence of CR or CRh to the date of first documented disease relapse or death. DOCRh is only defined for participants who achieve a CR or CRh.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR will be calculated as the date of the first response to the date of first documented disease relapse, disease progression, or death. DOR is only defined for participants who achieve a CR, CRi (including CRp), PR, and/or MLFS.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

10. Secondary Outcome: Duration of CRi (DOCRi)
Description: DOCRi will be calculated as the date of the first occurrence of CR or CRi (including CRp) to the date of the first documented relapse or death. DOCRi is only defined for participants who achieve a CR or CRi (including CRp).
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

11. Secondary Outcome: Time to CR (TTCR)
Description: TTCR will be assessed from the date of randomization to the date of first occurrence of CR. TTCR is only defined for participants who achieve a CR.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

12. Secondary Outcome: Time to CRh (TTCRh)
Description: TTCRh will be assessed from the date of randomization to the date of first occurrence of CR or CRh. TTCRh is only defined for participants who achieve a CR or CRh.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

13. Secondary Outcome: Time to Response (TTR)
Description: TTR will be assessed from the date of randomization to the date of the first response. TTR is only defined for participants who achieve a CR, CRi (including CRp), PR, and/or MLFS.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Time to CRi (TTCRi)
Description: TTCRi will be assessed from the date of randomization to the date of first occurrence of CR or CRi (including CRp). TTCRi is only defined for participants who achieve a CR or CRi (including CRp).
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

15. Secondary Outcome: Percentage of Participants With Abnormalities in Vital Sign Measurements
Description: Vital signs will include body temperature, respiratory rate, blood pressure, and heart rate.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

16. Secondary Outcome: Percentage of Participants With Abnormalities in Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

17. Secondary Outcome: Percentage of Participants With Abnormalities in 12-lead Electrocardiograms (ECGs)
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

18. Secondary Outcome: Percentage of Participants With Abnormalities in Echocardiogram (ECHO) or Multi-Gated Acquisition (MUGA) for Left Ventricular Ejection Fraction (LVEF)
Description: LVEF is determined by ECHO or MUGA scan in participants.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

19. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Tests
Description: Clinical laboratory assessments will include hematology, serum chemistry, coagulation.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

20. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered an investigational medicinal product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

21. Secondary Outcome: Percentage of Participants With AEs of Special Interest (AESIs)
Description: AESIs are AEs that are not solicited local or systemic AEs, they are predefined AEs that required close monitoring and prompt reporting to the sponsor. AESIs include protocol-specified QT prolongation, isocitrate dehydrogenase (IDH) differentiation syndrome and leukocytosis.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

22. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

23. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation or Death
Description: as for outcome 20
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

24. Secondary Outcome: Percentage of Participants Using Concomitant Medications
Description: Participants receiving concomitant medications will be adequately monitored by ECG controls, drug concentration (where applicable), and serum electrolytes (i.e., potassium and magnesium).
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

25. Secondary Outcome: Units of Platelets and Red Blood Cells (RBC) Infused
Description: All measures that are indicative of clinical benefit are measured like number of units of platelet and RBC infused.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

26. Secondary Outcome: Rate of Infection
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

27. Secondary Outcome: Number of Days Spent Hospitalized
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

28. Secondary Outcome: Change From Baseline in the European Organisation for Research and Treatment of Cancer (EORTC) QLC-C30 Questionnaire
Description: The EORTC QLQ-C30 questionnaire measures quality of life and consists of 30 questions that are incorporated into 5 functional domains (physical, role, cognitive, emotional, and social); a global health status/global quality of life; 3 symptom scales (fatigue, pain, and nausea and vomiting); and 6 single items that assess additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and the perceived financial burden of treatment experienced by participants with cancer.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

29. Secondary Outcome: Change From Baseline in the EORTC EQ-5D-5L Questionnaire
Description: The EORTC EQ-5D-5L questionnaire measures quality of life and spans 5 dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, which are used to build a composite of the participant's health status.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

30. Secondary Outcome: Percentage of Participants With CR With IDH1 Mutation Clearance (MC)
Description: CR with IDH1 MC is defined as a response of CR where there is no evidence of the IDH1 mutation by molecular techniques to below the level of detection (0.02%-0.04%) for ≥1 on-treatment time point. A CMH test will be used to compare the rate of CR between 2 treatment arms.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

31. Secondary Outcome: Percentage of Participants With Drug Exposure, Dose Modifications and Dose Intensities
Description: The number of doses administered, total dose, duration of treatment, dose intensity, and the proportion of participants with dose modifications, will be summarized by treatment arm.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

32. Secondary Outcome: Circulating Plasma Concentration of AG-120
Description: Serial blood samples will be drawn before and after dosing of study treatment in order to determine circulating plasma concentrations.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

33. Secondary Outcome: Circulating Plasma Concentration of 2-HG
Description: as for outcome 32
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: 3 years
Description: SAS included all participants who received at least 1 dose of the study treatment.
Arm/Group | AG-120 + Azacitidine | Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 27/71 | 45/73
Serious Adverse Events (participants affected / at risk) | 49/71 | 60/73
Other Adverse Events (participants affected / at risk) | 68/71 | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-120 + Azacitidine (N=71) | Placebo + Azacitidine (N=73)
Pneumonia (Infections and infestations) | 14 | 16
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 2
COVID-19 (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 2
Aspergillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Corynebacterium sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Enterococcal sepsis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pyrexia (General disorders) | 4 | 3
Fatigue (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Blast cell count increased (Investigations) | 1 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-120 + Azacitidine (N=71) | Placebo + Azacitidine (N=73)
Anaemia (Blood and lymphatic system disorders) | 22 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 9
Leukocytosis (Blood and lymphatic system disorders) | 8 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 20 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 14
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Constipation (Gastrointestinal disorders) | 19 | 38
Diarrhoea (Gastrointestinal disorders) | 25 | 25
Haemorrhoids (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 30 | 28
Proctalgia (Gastrointestinal disorders) | 1 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 28 | 19
Asthenia (General disorders) | 11 | 24
Chest discomfort (General disorders) | 2 | 4
Fatigue (General disorders) | 9 | 10
Injection site reaction (General disorders) | 4 | 5
Non-cardiac chest pain (General disorders) | 4 | 2
Oedema peripheral (General disorders) | 8 | 16
Pyrexia (General disorders) | 23 | 29
Oral candidiasis (Infections and infestations) | 1 | 5
Oral herpes (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 8 | 9
Suspected COVID-19 (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 7
Fall (Injury, poisoning and procedural complications) | 3 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 4 | 3
C-reactive protein increased (Investigations) | 3 | 4
Electrocardiogram QT prolonged (Investigations) | 14 | 5
Neutrophil count decreased (Investigations) | 6 | 5
Platelet count decreased (Investigations) | 8 | 6
Weight decreased (Investigations) | 4 | 11
Decreased appetite (Metabolism and nutrition disorders) | 11 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Dizziness (Nervous system disorders) | 7 | 3
Dysgeusia (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 8 | 2
Syncope (Nervous system disorders) | 5 | 4
Anxiety (Psychiatric disorders) | 5 | 3
Confusional state (Psychiatric disorders) | 5 | 5
Delirium (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 13 | 9
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Erythema (Skin and subcutaneous tissue disorders) | 6 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Haematoma (Vascular disorders) | 9 | 1
Hypertension (Vascular disorders) | 7 | 4
Hypotension (Vascular disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03173248/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03173248/SAP_001.pdf